CLINICAL TRIAL: NCT03593707
Title: A PHASE 1, RANDOMIZED, OPEN-LABEL, TWO-PERIOD, TWO-SEQUENCE, CROSSOVER STUDY TO EVALUATE THE EFFECT OF PF-06865571 ON THE PHARMACOKINETICS OF METFORMIN IN HEALTHY ADULT SUBJECTS
Brief Title: Drug-Drug Interaction Study to Evaluate the Effect of PF-06865571 on Metformin Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: C2541006; 2018-001888-23 (EudraCT Number)
Record Dates: First submitted 2018-07-10; First posted 2018-07-20 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Healthy Volunteers
Keywords: PF-06865571; Metformin; Drug-drug interaction; Pharmacokinetics
MeSH Terms: interventions — Metformin; ervogastat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Metformin Alone (Experimental): Metformin alone
  Interventions: Drug: Metformin
- Metformin + PF-06865571 (Experimental): Co-administer metformin and PF-06865571
  Interventions: Drug: Metformin; Drug: PF-06865571

INTERVENTIONS:
Drug: Metformin — Metformin
  Other Names: Glucophage
Drug: PF-06865571 — PF-06865571
  Arms: Metformin + PF-06865571

SUMMARY:
This study is designed to assess the effect of PF-06865571 administration on the pharmacokinetics of metformin in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female subjects of nonchildbearing potential and/or male subjects who, at the time of screening, are between the ages of 18 and 55 years.
2. Body mass index of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).
3. Evidence of a personally signed and dated informed consent document.
4. Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. Any condition possibly affecting drug absorption (eg, gastrectomy).
3. A positive urine drug test.
4. History of regular alcohol consumption exceeding 14 drinks/week for female subjects or 21 drinks/week for male subjects.
5. Treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of investigational product (whichever is longer).
6. Screening supine BP >=140 mm Hg (systolic) or >=90 mm Hg (diastolic), following at least 5 minutes of supine rest.
7. Screening supine 12-lead ECG demonstrating a corrected QT (QTc) interval >450 msec or a QRS interval >120 msec.
8. Subjects with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study-specific laboratory and confirmed by a single repeat test, if deemed necessary:

   * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level >=1.25× upper limit of normal (ULN);
   * Total bilirubin level >=1.5× ULN; subjects with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is <=ULN.
9. Fertile male subjects who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and through the follow up contact, or have female partners that are pregnant.
10. Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of investigational product.
11. Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
12. History of sensitivity to heparin or heparin-induced thrombocytopenia only if heparin is used to flush any intravenous catheters in the study.
13. History of human immunodeficiency virus (HIV), hepatitis B, or hepatitis C; positive testing at the screening visit for HIV, hepatitis B surface antigen (HepBsAg), hepatitis B core antibody (HepBcAb), or hepatitis C antibody (HCVAb). While not part of the tests assessed in this study, subjects with a positive hepatitis B surface antibody (HepBsAb) result due to vaccination are deemed eligible.
14. Unwilling or unable to comply with the criteria in the Lifestyle Requirements section of this protocol.
15. Subjects who are investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or subjects who are Pfizer employees, including their family members, directly involved in the conduct of the study.
16. Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
17. Subjects who have participated in prior studies with PF-06865571.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2018-08-17 (Actual); Primary Completion 2019-01-17 (Actual); Study Completion 2019-02-13 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Metformin (in absence of PF-06865571) | 0, 0.5, 1, 2, 4, 6, 8, 10, 12, 16, 24, 48 hours post-dose
  Metformin Cmax in absence of PF-06865571
Metformin Cmax (in presence of PF-06865571) | 0, 0.5, 1, 2, 4, 6, 8, 10, 12, 16, 24, 48 hours post-dose
  Metformin Cmax in presence of PF-06865571
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) of Metformin (in absence of PF-06865571) | 0, 0.5, 1, 2, 4, 6, 8, 10, 12, 16, 24, 48 hours post-dose
  Metformin AUCinf in absence of PF-06865571
Metformin AUCinf (in presence of PF-06865571) | 0, 0.5, 1, 2, 4, 6, 8, 10, 12, 16, 24, 48 hours post-dose
  Metformin AUCinf in presence of PF-06865571

SECONDARY OUTCOMES:
Number of Participants With Treatment Emergent Treatment-Related Adverse Events (AEs) | Baseline up to 35 days after last dose of study medication
  Treatment-related AE are any untoward medical occurrence attributed to study drug in a participant who received study drug. Treatment-emergent are events between first dose of study drug and up to 35 days after last dose that were absent before treatment or that worsened relative to pretreatment state. Relatedness to study drug is assessed either yes or no by the investigator. Participants with multiple occurrences of an AE within a category are counted once within the category.
Number of Participants With Laboratory Abnormalities | Baseline up to 35 days after last dose of study medication
  The following parameters were analyzed for laboratory examination: hematology (hemoglobin, hematocrit, red blood cell count, platelet count, white blood cell count, total neutrophils, eosinophils, monocytes, basophils, lymphocytes); blood chemistry (blood urea nitrogen, creatinine, glucose, calcium, sodium, potassium, chloride, total bicarbonate, aspartate aminotransferase, alanine aminotransferase, total bilirubin, alkaline phosphatase, uric acid albumin, total protein); urinalysis (decimal logarithm of reciprocal of hydrogen ion activity [pH], glucose, protein, blood, ketones, microscopy [if urine tested positive for blood or protein]).
Number of Participants With Clinically Significant Change From Baseline in Vital Signs | 0 and 48 hours (h) post-dose
  the following parameters were analyzed for examination of vital signs: systolic and diastolic blood pressure and pulse rate.
Number of Participants With Change From Baseline in Electrocardiogram (ECG) Findings | 0 and 48 h post-dose
  Absolute values and changes from baseline for ECG parameters

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=C2541006&StudyName=A+Phase+1%2C+Randomized%2C+Open-label%2C+Two-period%2C+Two-sequence%2C+Crossover+Study+To+Evaluate+The+Effect+Of+Pf-06865571+On+The+Pharmacokinetics+Of+Metformin+In+Healthy+Adult+Subjects